CLINICAL TRIAL: NCT05806619
Title: Glioma: BIOMOLECULAR Aspects From Tissue to Radiomics
Brief Title: Glioma: Biomolecular Aspects
Acronym: GLIOMA
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1271/19
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected glioma: Patients at diagnosis of both sexes with suspected glioma
  Interventions: Other: histopathological analysis; morphological and non-morphological magnetic resonance
- Patients at relapse/progression: Patients at relapse/progression with neurosurgical reoperation indication
  Interventions: Other: histopathological analysis; morphological and non-morphological magnetic resonance

INTERVENTIONS:
Other: histopathological analysis; morphological and non-morphological magnetic resonance — The surgical material removed during surgery was subjected to histological analysis. Morphological and non-morphological magnetic resonance examination before the neurosurgical surgery, according to clinical practice.

SUMMARY:
Main limitations in Glioma studies are due to the wide heterogeneity and genetic instability of the tumor and to the fact that the molecular informations are static, i.e. obtained on the tumor at its onset. Instead, spontaneous or therapy-induced variations are difficult to evaluate and they would need further sampling of the tumor throughout the clinical history. Currently these data are more and more routinely used not only for diagnostics but also in the clinical management of the patient.

Furthermore, microenvironment study is becoming increasingly important. It is also important correlate morpho-functional pathway and brain Magnetic Resonance.

Therefore, the main goal of the study is to correlate the data obtained with morphological (site, signal intensity, margins, behavior after contrast medium infusion, mismatch between T2 and FLAIR sequences) and non-morphological MR imaging through a radiomic approach and Diffusion and Perfusion study, with molecular data relating to the IDH mutation, MGMT gene promoter methylation, 1p/19q co-deletion and EGFRvIII expression.

Furthermore, it is proposed to carry out a correlation between the radiological data and the mutations found in the NGS panel.

ELIGIBILITY:
Inclusion Criteria:

* glioma diagnosis
* have performed morphological brain MRI or not with contrast medium before surgery
* informed consent form

Exclusion Criteria:

* Patients without Magnetic Resonance were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected glioma who have been subjected to surgery at diagnosis or recurrence
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between MR and molecular data | 24 months
  Demonstrate the existence of a correlation between the non-morphological brain Magnetic Resonance (MR) data obtained with diffusion and perfusion techniques and molecular data, in particular with MGMT gene methylation.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - San Giovanni Addolorata Hospital, Rome, Roma
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided